CLINICAL TRIAL: NCT02496793
Title: A Community Randomized Study to Evaluate the Effect of a Community-Based Peer Facilitator Intervention on Prevention of Maternal to Child Transmission (PMTCT) of HIV Program Outcomes in Zimbabwe
Brief Title: Community-Based Peer Facilitator Intervention (Zimbabwe)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Ministry of Health and Child Welfare, Zimbabwe (Other); The Children's Investment Fund Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EG0090; MRCZ/A/1651 (Other: Medical Research Council of Zimbabwe)
Record Dates: First submitted 2015-06-24; First posted 2015-07-14 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: HIV-infection/Aids
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer Facilitator and Support Group (Experimental): Peer-facilitated community support group is the experimental intervention. The intervention tested in this study involved using trained peer facilitators to create demand for and retention within the ANC/PMTCT program.The peer facilitators were volunteer women from the community, who had recently been through the ANC process themselves and could speak about their experience(s). the support group meetings was to develop skills and generate self-efficacy for the women to be able to take actions such as routine antenatal and postnatal clinic attendance using participatory learning techniques. The peer facilitators were provided with job aids which outlined key points for the various educational sessions.
  Interventions: Behavioral: Peer-facilitated community support group
- Standard Care (No Intervention): ANC/PMTCT activities as per standard of care in Zimbabwe

INTERVENTIONS:
Behavioral: Peer-facilitated community support group — Support groups were composed of up to 20 women from community. Peer facilitator facilitated a total of 6 groups of a maximum of 20 women each. Women were exposed to 8 two hour sessions. Facilitators gave activities in support of MCH/PMTCT. Group met twice a month for four months. The support group meetings took place in the community at a convenient location for those attending (e.g. village meeting point, churches, schools or individual households). With local support through community leaders, the intervention involved trained peer facilitators working with pregnant and post-partum women to form ANC and PNC support groups through which they will present information on general maternal and child health and PMTCT specific topics using participatory learning and problem-solving approaches.
  Arms: Peer Facilitator and Support Group

SUMMARY:
The goal of this community randomized operations research study was to evaluate the effect of a peer-facilitated community support group intervention on uptake of maternal and neonatal child health (MNCH) and PMTCT services and on adherence outcomes in Zimbabwe.

DETAILED DESCRIPTION:
To increase uptake of, and retention within maternal and child health/prevention of maternal-to-child HIV transmission (MCH/PMTCT) services, the investigators conducted a community-based peer facilitator intervention study in Hurungwe District of Zimbabwe. Using a paired community randomized design, 16 health facility-linked communities were randomly allocated to the intervention or control condition, with a total of approximately 1,600 pregnant and lactating women, (100 women in each community), recruited into the study. In the intervention communities, 24 trained peer facilitators (3 in each community) using participatory educational approaches were encouraging women to form antenatal and post-natal groups, and to utilize and adhere to MCH/PMTCT services and recommendations.

Peer facilitators, by the definition of this project, were women from the community who were peers to pregnant and lactating women; who had recently been through the process themselves and could speak to their experience. A key activity of the community-based peer facilitators was the encouragement of the formation of women into groups, and the participation of these women into antenatal care (ANC), prevention of maternal to child transmission (PMTCT), and postnatal care (PNC) programs. The group process was enable solidarity and support among the women at the vulnerable times of pregnancy and lactation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and breastfeeding women who were 18 years of age and above, regardless of HIV status, were eligible to participate in support groups.

Exclusion Criteria:

* Women less than 18 years and those who were mentally ill were excluded as they could not give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To measure proportion of women less than 20 weeks gestation at first ANC attendance | 12 months
  The number of women attending first ANC attendance at 20 weeks gestation as a proportion of all women attending first ANC attendance at any age of gestation
To measure proportion of pregnant women attending four ANC visits | 12 months
  The number of pregnant women attending four ANC visits as a proportion of pregnant women attending any ANC visit
To measure proportion of HIV exposed babies tested for HIV | 12 months
  The number of HIV exposed babies test for HIV as a proportion of the number of HIV exposed babies
To measure proportion of HIV exposed babies initiated on NVP prophylaxis at birth | 12 months
  The number of HIV exposed babies initiated on NVP prophylaxis at birth as a proportion of the number of HIV exposed babies tested for HIV at birth

SECONDARY OUTCOMES:
Pregnant and postnatal women tested for HIV as a proportion of these women in the community | 12 months
  The number of pregnant and postnatal women tested for HIV as a proportion of the number of pregnant and postnatal women estimated to have HIV in the community

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey J Woelk, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation